CLINICAL TRIAL: NCT00740714
Title: Effects of Coenzyme Q10 in Parkinson Disease - Phase III
Brief Title: Effects of Coenzyme Q10 (CoQ) in Parkinson Disease
Acronym: QE3
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The investigational drug is unlikely to demonstrate efficacy over placebo for this indication. However, no safety issues were discovered.
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH); University of Rochester (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: U01NS050324 (NIH); U01NS050573 (NIH)
Record Dates: First submitted 2008-08-22; First posted 2008-08-25 (Estimated); Results first posted 2013-01-31 (Estimated); Last update posted 2013-01-31 (Estimated); Status verified 2012-12

CONDITIONS: Parkinson Disease
Keywords: Parkinson disease; PD; Coenzyme Q10; CoQ
MeSH Terms: conditions — Parkinson Disease | interventions — coenzyme Q10; Vitamin E; Ubiquinone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- A (Experimental): Randomized to active treatment (Coenzyme Q10 2400 mg/day with vitamin E 1200 IU/day)
  Interventions: Drug: Coenzyme Q10 with vitamin E
- B (Experimental): Randomized to active treatment (Coenzyme Q10 1200 mg/day with vitamin E 1200 IU/day)
  Interventions: Drug: Coenzyme Q10 with vitamin E
- C (Placebo Comparator): Placebo (with vitamin E 1200 IU/day)
  Interventions: Drug: placebo with vitamin E

INTERVENTIONS:
Drug: Coenzyme Q10 with vitamin E — 2400 mg dose - eight 300 mg Coenzyme Q10 chewable wafers taken orally four times a day; 1200 mg dose - four 300 mg Coenzyme Q10 and four placebo chewable wafers taken orally four times a day.
  Other Names: Coenzyme Q10, ubiquinone, ubidecarenone
  Arms: A; B
Drug: placebo with vitamin E — placebo or an inactive substance (with vitamin E 1200 IU/day); Placebo - eight chewable wafers taken orally four times a day.
  Arms: C

SUMMARY:
The purpose of this study is to evaluate the safety and effectiveness of high dosages of Coenzyme Q10 in slowing clinical decline in people who have early Parkinson disease.

DETAILED DESCRIPTION:
Parkinson disease (PD) is a progressive neurodegenerative disease that affects more than 1,000,000 Americans. Currently there is no proven therapy to reduce the rate of progression of PD. In a previous phase II clinical trial, investigators demonstrated that Coenzyme Q10 (CoQ) at dosages of 300, 600, and 1200 mg/day was safe and well-tolerated in individuals with early, untreated PD. The findings also suggested that CoQ may slow the progressive impairment of PD as measured by the Unified Parkinson Disease Rating Scale (UPDRS).

In this study, researchers will conduct a randomized, placebo-controlled, phase III trial of CoQ to confirm and extend the results of the earlier phase II study. The primary objective of this trial is to compare the effect of two dosages of CoQ (1200 and 2400 mg/day) and placebo on the total UPDRS score in people with early PD. The study also will evaluate independent function, cognition, and quality of life. Plasma CoQ levels will be measured at months 1, 8 and 16 and correlated with changes in UPDRS scores.

Participants will be randomly assigned to receive a placebo (an inactive substance), 1200 mg/d CoQ, or 2400 mg/d CoQ. They will be evaluated at screening, baseline, and during visits at months 1, 4, 8, 12, and 16. Information gained from this trial could lead to changes in management of people with early PD.

ELIGIBILITY:
Inclusion Criteria:

* Presence of all 3 of the cardinal features of Parkinson disease (resting tremor, bradykinesia and rigidity). The clinical signs must be asymmetric.
* The diagnosis of Parkinson disease within 5 years prior to the Screening Visit.
* Age 30 or older.
* Female subjects must not be of childbearing potential or must use an approved form of contraception for the duration of the trial.

Exclusion Criteria:

* Use of any Parkinson disease medication within 60 days prior to the Baseline Visit.
* Duration of previous use of symptomatic medication for Parkinson disease cannot exceed 90 days such as levodopa, dopaminergic agonists (including ropinirole, pramipexole, pergolide, cabergoline, and the rotigotine transdermal system), selegiline, rasagiline, amantadine, and anticholinergic agents.
* Parkinsonism due to drugs including neuroleptics, alphamethyldopa, reserpine, metoclopramide, valproic acid.
* Use of antioxidants (such as selegiline, rasagiline, vitamins E and C), additional supplemental vitamins or minerals, regular use of neuroleptics, chloramphenicol, valproic acid, warfarin.
* Other parkinsonian disorders.
* Modified Hoehn and Yahr score of 3 or greater at Screening Visit or Baseline Visit.
* UPDRS tremor score of 3 or greater at Screening Visit or Baseline Visit.
* Mini-Mental State Examination (MMSE) score of 25 or less.
* History of stroke.
* Disability sufficient to require treatment with dopaminergic medication or anticipated need for dopaminergic medication within next 3 months.
* Other serious illness, including psychiatric illness.
* Patients with active cardiovascular, peripheral vascular or cerebrovascular disease within the past year.
* Clinically serious abnormalities in the Screening Visit laboratory studies or electrocardiogram.
* Use of methylphenidate, cinnarizine, reserpine, amphetamine or a MAO-A inhibitor within 6 months prior to the Baseline Visit.
* Unstable dose of CNS active therapies.
* Use of appetite suppressants within 60 days prior to the Baseline Visit.
* History of active epilepsy within the last 5 years.
* Revised Hamilton Rating Scale for Depression of 11 or greater.
* Participation in other drug studies or use of other investigational drugs within 30 days prior to Screening Visit.
* History of electroconvulsive therapy.
* History of any brain surgery for Parkinson disease.
* History of structural brain disease such as prior trauma causing damage detected on a CT scan or MRI, hydrocephalus, or prior brain neoplasms.

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Actual)
Dates: Start 2008-12; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: M. Flint Beal, MD, Principal Investigator — Weill Medical College of Cornell University, New York Hospital Department of Neurology; David Oakes, PhD, Principal Investigator — University of Rochester, Department of Biostatistics; Ira Shoulson, MD, Principal Investigator — University of Rochester, Clinical Trials Coordination Center
Locations (68):
- United States (59):
  - University of Alabama, Birmingham, 350 Sparks Center, 1720 7Th Avenue South, Birmingham, Alabama
  - Barrow Neurological Clinics At St Joseph'S Hospital & Medical Center, 500 West Thomas Road Suite 720, Phoenix, Arizona
  - Mayo Clinic Arizona, 13400 East Shea Boulevard, Desk 34 3B, Scottsdale, Arizona
  - Sunhealth Research Institute, 10515 West Santa Fe Drive, Sun City, Arizona
  - The Parkinson'S & Movement Disorder Institute, 9940 Talbert Avenue, Suite 204, Fountain Valley, California
  - University of California Irvine, 100 Irvine Hall, Irvine, California
  - University of California San Diego, Alzheimer'S Disease Research Center, 9500 Gilman Drive, La Jolla, California
  - UCLA Medical Center, 710 Westwood Plaza, A-253, Los Angeles, California
  - UC Davis Dept of Neurology, 4860 Y Street, Suite 3700, Sacramento, California
  - The Parkinson's Institute, 675 ALMANOR AVENUE, Sunnyvale, California
  - Department of Neurology/Mail Stop B185, 12631 East 17Th Avenue Room 5209, Academic Office 1 Po Box 6511, Aurora, Colorado
  - Colorado Neurological Institute, 701 East Hampden Avenue, Suite 510, Littleton, Colorado
  - The Institute For Neurodegenerative Disorders, 60 Temple Street, Suite 8B, New Haven, Connecticut
  - University of Florida, McKnight Brain Institute Po Box 100236, 100 S Newell Drive L3-100, Gainsville, Florida
  - University of Miami, 1501 North West 9Th Avenue Second Floor, Department of Neurology D4-5, Miami, Florida
  - University of South Florida, 4 Columbia Drive, Suite 410, Tampa, Florida
  - Emory University School of Medicine, Wesley Woods Health Center, 1841 Clifton Road NE Room 328, Atlanta, Georgia
  - Movement Disorders Program, Department of Neurology, Medical College of Georgia, Augusta, Georgia
  - Northwestern University, 710 North Lake Shore Drive, Chicago, Illinois
  - Rush University Medical Center Department of Neurological Sciences, 1725 West Harrison Suite 755, Chicago, Illinois
  - University of Chicago, 5841 South Maryland Avenue, Mc2030, Chicago, Illinois
  - Indiana University School of Medicine, Outpatient Clinical Research Facility, 535 Barnhill Drive Room #150, Indianapolis, Indiana
  - University of Iowa Hospitals, 2133 Rcp Department of Neurology, 200 Hawkins Drive, Iowa City, Iowa
  - The University of Kansas Medical Center, Department of Neurology Ms #2012, 3599 Rainbow Boulevard, Kansas City, Kansas
  - University of Louisville, Movement Disorder Clinic, Frazier Rehab, 220 Abraham Flexner, Suite 606, Louisville, Kentucky
  - Ochsner Clinic Foundation, 1514 Jefferson Highway, Dept of Neurology 7Th Floor, New Orleans, Louisiana
  - Lsuhsc Shreveport, Department of Neurology, 1501 Kings Highway Room 3-436, Shreveport, Louisiana
  - University of Maryland School of Medicine, 22 South Greene Street, N4 W49-B, Baltimore, Maryland
  - Johns Hopkins, 601 North Caroline Street, Suite 5064, Baltimore, Maryland
  - Parkinson & Movement Dis Center If Maryland, 8180 Lark Brown Road, Suite 101, Elkridge, Maryland
  - Boston University Medical Center, Department of Neurology, 715 Albany Street C329, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, 330 Brookline Avenue, Shapiro 809D, Boston, Massachusetts
  - University of Minnesota, 420 Delaware Street SE, Mmc 295, Minneapolis, Minnesota
  - Washington University School of Medicine, 660 South Euclid, Box 8111, St Louis, Missouri
  - Albany Medical College, Parkinson'S Disease & Movement Disorders Ctr, 47 New Scottland Avenue, Albany, New York
  - Suny Downstate Medical Center , 450 Clarkson Avenue , Box 1213, Brooklyn, New York
  - Northshore-Lij Health System, the Feinstein Institute Fpr Medical Research, 350 Community Drive Room 100, Manhasset, New York
  - Beth Israel Medical Center, 10 Union Square East, Suite 5Hh2, New York, New York
  - Beth Israel Medical Center, Phillips Ambulatory Care Center, 10 Union Square East Room 5Ho1, New York, New York
  - Parkinson'S Dis & Movement Disorders Inst, 428 East 72Nd Street, Suite 400, New York, New York
  - Weill Medical College of Cornell, New York, New York
  - Columbia University, 710 West 168Th Street, 3Rd Floor, New York, New York
  - University of Rochester Department of Neurology, 919 Westfall Road Building C Suite 220, Rochester, New York
  - JACOBI MEDICAL CENTER, 1400 Pelham Pkwy S, The Bronx, New York
  - Duke University Medical Center, Duke Health Center At Morreene Road, 932 Morreene Road Room 213, Durham, North Carolina
  - University Neurology Inc., 222 Piedmont Avenue, Suite 3200, Cincinnati, Ohio
  - The Cleveland Clinic Foundation, 9500 Euclid Avenue S-31, Cleveland, Ohio
  - Ohio State University Medical Center, 1581 Dodd Drive, 371 McCampbell Hall, Columbus, Ohio
  - University of Toledo , 3000 Arlington Avenue , Mail Stop 1195, Toledo, Ohio
  - Oregon Health & Science University, Dept of Neurology, 3181 SW Sam Jackson Park Road Op-32, Portland, Oregon
  - Penn State Milton S Hershey Med Center, Department of Neurology Mc H109 Room 2846, 500 University Drive Po Box 850, Hershey, Pennsylvania
  - University of Pennsylvania, Pennsylvania Hospital Department of Neurology, 330 South 9Th Street, Philadelphia, Pennsylvania
  - Neurohealth Parkinson'S Disease, Movement Disorder Center, 227 Centerville Road, Warwick, Rhode Island
  - Medical University of South Carolina, Charleston Memorial Hospital, 326 Calhoun Street Suite 308, Charleston, South Carolina
  - Semmes Murphey Clinic, 1211 Union Avenue, Suite 200, Memphis, Tennessee
  - Baylor College of Medicine - Parkinson'S, Disease Center and Movement Disorders Clinic, 65501 Fannin St, Suite 1801, Houston, Texas
  - University of Vermont , Department of Neurology Given Building C-219 , 89 Beaumont Avenue, Burlington, Vermont
  - Booth Gardner Parkinson'S Care Center, 13030 121St Way North East Suite 203, Kirkland, Washington
  - Medical College of Wisconsin, Department of Neurology, 9200 West Wisconsin Avenue, Milwaukee, Wisconsin
- Canada (9):
  - Un of Calgary Movement Disorders Program, Dept of Clin Neurosciences Area 3 Neurology, 3350 Hospital Dr NW Health Sciences Centre, Calgary, Alberta
  - University of Alberta Glenrose Rehab Hosp, Rm 0601 Glen East, 10230 - 111 Avenue, Edmonton, Alberta
  - London Health Sciences Centre, University Campus Room 10N29, 339 Windermere Road, London, Ontario
  - The Ottawa Hospital-Civic Campus, 1053 Carling Avenue C2 Room 2210, Ottawa, Ontario
  - Toronto Western Hospital, Univ Health Network, 399 Bathurst Street Mc 7-402, Movement Disorders Centre, Toronto, Ontario
  - CHUM-HOPITAL NOTRE DAME, 1560 rue SHERBROOKE est ROOM GR 1185, PAVILLON DECHAMPS etage rez-de-chaussee, Montreal, Quebec
  - Quebec Memory and Motor Skills Dis Clinic, Price Building 3Rd Floor, 65 Sainte-Anne Street, Québec, Quebec
  - University of Sherbrooke, 3001 12E Avenue Nord, Sherbrooke, Quebec
  - Royal University Hospital, 103 Hospital Drive, Room 1663, Saskatoon, Saskatchewan

REFERENCES:
- [Background] Beal MF, Henshaw DR, Jenkins BG, Rosen BR, Schulz JB. Coenzyme Q10 and nicotinamide block striatal lesions produced by the mitochondrial toxin malonate. Ann Neurol. 1994 Dec;36(6):882-8. doi: 10.1002/ana.410360613. PMID 7998775
- [Background] Beal MF, Matthews RT, Tieleman A, Shults CW. Coenzyme Q10 attenuates the 1-methyl-4-phenyl-1,2,3,tetrahydropyridine (MPTP) induced loss of striatal dopamine and dopaminergic axons in aged mice. Brain Res. 1998 Feb 2;783(1):109-14. doi: 10.1016/s0006-8993(97)01192-x. PMID 9479058
- [Background] Beal MF. Energetics in the pathogenesis of neurodegenerative diseases. Trends Neurosci. 2000 Jul;23(7):298-304. doi: 10.1016/s0166-2236(00)01584-8. PMID 10856939
- [Background] Beal MF. Coenzyme Q10 as a possible treatment for neurodegenerative diseases. Free Radic Res. 2002 Apr;36(4):455-60. doi: 10.1080/10715760290021315. PMID 12069110
- [Background] NINDS NET-PD Investigators. A randomized clinical trial of coenzyme Q10 and GPI-1485 in early Parkinson disease. Neurology. 2007 Jan 2;68(1):20-8. doi: 10.1212/01.wnl.0000250355.28474.8e. PMID 17200487
- [Background] Ravina BM, Fagan SC, Hart RG, Hovinga CA, Murphy DD, Dawson TM, Marler JR. Neuroprotective agents for clinical trials in Parkinson's disease: a systematic assessment. Neurology. 2003 Apr 22;60(8):1234-40. doi: 10.1212/01.wnl.0000058760.13152.1a. PMID 12707423
- [Background] Shoulson I, Oakes D, Fahn S, Lang A, Langston JW, LeWitt P, Olanow CW, Penney JB, Tanner C, Kieburtz K, Rudolph A; Parkinson Study Group. Impact of sustained deprenyl (selegiline) in levodopa-treated Parkinson's disease: a randomized placebo-controlled extension of the deprenyl and tocopherol antioxidative therapy of parkinsonism trial. Ann Neurol. 2002 May;51(5):604-12. doi: 10.1002/ana.10191. PMID 12112107
- [Background] Shults CW, Haas RH, Passov D, Beal MF. Coenzyme Q10 levels correlate with the activities of complexes I and II/III in mitochondria from parkinsonian and nonparkinsonian subjects. Ann Neurol. 1997 Aug;42(2):261-4. doi: 10.1002/ana.410420221. PMID 9266740
- [Background] Shults CW, Beal MF, Fontaine D, Nakano K, Haas RH. Absorption, tolerability, and effects on mitochondrial activity of oral coenzyme Q10 in parkinsonian patients. Neurology. 1998 Mar;50(3):793-5. doi: 10.1212/wnl.50.3.793. PMID 9521279
- [Background] Shults CW, Oakes D, Kieburtz K, Beal MF, Haas R, Plumb S, Juncos JL, Nutt J, Shoulson I, Carter J, Kompoliti K, Perlmutter JS, Reich S, Stern M, Watts RL, Kurlan R, Molho E, Harrison M, Lew M; Parkinson Study Group. Effects of coenzyme Q10 in early Parkinson disease: evidence of slowing of the functional decline. Arch Neurol. 2002 Oct;59(10):1541-50. doi: 10.1001/archneur.59.10.1541. PMID 12374491
- [Background] Shults CW. Coenzyme Q10 in neurodegenerative diseases. Curr Med Chem. 2003 Oct;10(19):1917-21. doi: 10.2174/0929867033456882. PMID 12871093
- [Background] Shults CW, Flint Beal M, Song D, Fontaine D. Pilot trial of high dosages of coenzyme Q10 in patients with Parkinson's disease. Exp Neurol. 2004 Aug;188(2):491-4. doi: 10.1016/j.expneurol.2004.05.003. PMID 15246848
- [Background] Lee IM, Cook NR, Gaziano JM, Gordon D, Ridker PM, Manson JE, Hennekens CH, Buring JE. Vitamin E in the primary prevention of cardiovascular disease and cancer: the Women's Health Study: a randomized controlled trial. JAMA. 2005 Jul 6;294(1):56-65. doi: 10.1001/jama.294.1.56. PMID 15998891
- [Background] Blatt DH, Pryor WA. High-dosage vitamin E supplementation and all-cause mortality. Ann Intern Med. 2005 Jul 19;143(2):150-1; author reply 156-8. doi: 10.7326/0003-4819-143-2-200507190-00018. No abstract available. PMID 16027460
- [Background] McDonald SR, Sohal RS, Forster MJ. Concurrent administration of coenzyme Q10 and alpha-tocopherol improves learning in aged mice. Free Radic Biol Med. 2005 Mar 15;38(6):729-36. doi: 10.1016/j.freeradbiomed.2004.11.014. PMID 15721983
- [Background] Miller ER 3rd, Pastor-Barriuso R, Dalal D, Riemersma RA, Appel LJ, Guallar E. Meta-analysis: high-dosage vitamin E supplementation may increase all-cause mortality. Ann Intern Med. 2005 Jan 4;142(1):37-46. doi: 10.7326/0003-4819-142-1-200501040-00110. Epub 2004 Nov 10. PMID 15537682
- [Background] Parkinson Study Group. Effects of tocopherol and deprenyl on the progression of disability in early Parkinson's disease. N Engl J Med. 1993 Jan 21;328(3):176-83. doi: 10.1056/NEJM199301213280305. PMID 8417384
- [Derived] Parkinson Study Group QE3 Investigators; Beal MF, Oakes D, Shoulson I, Henchcliffe C, Galpern WR, Haas R, Juncos JL, Nutt JG, Voss TS, Ravina B, Shults CM, Helles K, Snively V, Lew MF, Griebner B, Watts A, Gao S, Pourcher E, Bond L, Kompoliti K, Agarwal P, Sia C, Jog M, Cole L, Sultana M, Kurlan R, Richard I, Deeley C, Waters CH, Figueroa A, Arkun A, Brodsky M, Ondo WG, Hunter CB, Jimenez-Shahed J, Palao A, Miyasaki JM, So J, Tetrud J, Reys L, Smith K, Singer C, Blenke A, Russell DS, Cotto C, Friedman JH, Lannon M, Zhang L, Drasby E, Kumar R, Subramanian T, Ford DS, Grimes DA, Cote D, Conway J, Siderowf AD, Evatt ML, Sommerfeld B, Lieberman AN, Okun MS, Rodriguez RL, Merritt S, Swartz CL, Martin WR, King P, Stover N, Guthrie S, Watts RL, Ahmed A, Fernandez HH, Winters A, Mari Z, Dawson TM, Dunlop B, Feigin AS, Shannon B, Nirenberg MJ, Ogg M, Ellias SA, Thomas CA, Frei K, Bodis-Wollner I, Glazman S, Mayer T, Hauser RA, Pahwa R, Langhammer A, Ranawaya R, Derwent L, Sethi KD, Farrow B, Prakash R, Litvan I, Robinson A, Sahay A, Gartner M, Hinson VK, Markind S, Pelikan M, Perlmutter JS, Hartlein J, Molho E, Evans S, Adler CH, Duffy A, Lind M, Elmer L, Davis K, Spears J, Wilson S, Leehey MA, Hermanowicz N, Niswonger S, Shill HA, Obradov S, Rajput A, Cowper M, Lessig S, Song D, Fontaine D, Zadikoff C, Williams K, Blindauer KA, Bergholte J, Propsom CS, Stacy MA, Field J, Mihaila D, Chilton M, Uc EY, Sieren J, Simon DK, Kraics L, Silver A, Boyd JT, Hamill RW, Ingvoldstad C, Young J, Thomas K, Kostyk SK, Wojcieszek J, Pfeiffer RF, Panisset M, Beland M, Reich SG, Cines M, Zappala N, Rivest J, Zweig R, Lumina LP, Hilliard CL, Grill S, Kellermann M, Tuite P, Rolandelli S, Kang UJ, Young J, Rao J, Cook MM, Severt L, Boyar K. A randomized clinical trial of high-dosage coenzyme Q10 in early Parkinson disease: no evidence of benefit. JAMA Neurol. 2014 May;71(5):543-52. doi: 10.1001/jamaneurol.2014.131. PMID 24664227

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The recruitment period for the required 600 patients was from January 2009 to October 2010. There were 67 sites (60 in the US and 7 in Canada) that participated in the study. Most of these sites were located at or affiliated with large academic medical centers.
Pre-assignment Details: Patients were required to undergo a thorough screening visit. If patients were taking CoEnzyme Q10 but otherwise eligible for assignment, they were asked to return after a wash out period of 60 to 120 days based on daily dosage.
Groups:
- A. Coenzyme Q10 2400 mg/Day With Vitamin E 1200 IU/Day: Randomized to active treatment (Coenzyme Q10 2400 mg/day with vitamin E 1200 IU/day)
- B. Coenzyme Q10 1200 mg/Day With Vitamin E 1200 IU/Day: Randomized to active treatment (Coenzyme Q10 1200 mg/day with vitamin E 1200 IU/day)
- C. Placebo With Vitamin E 1200 IU/Day: Placebo (with vitamin E 1200 IU/day)
Period: Overall Study
Arm/Group | A. Coenzyme Q10 2400 mg/Day With Vitamin E 1200 IU/Day | B. Coenzyme Q10 1200 mg/Day With Vitamin E 1200 IU/Day | C. Placebo With Vitamin E 1200 IU/Day
Started | 196 (Randomized throughout the recruitment period) | 201 (Randomized throughout the recruitment period) | 203 (Randomized throughout the recruitment period)
Reaching Endpoint Before May 6, 2011 | 86 | 87 | 94
Active Patients at Study Termination | 24 | 12 | 33
Completed | 179 | 182 | 174
Not Completed | 17 | 19 | 29
Not completed — Withdrawal by Subject | 17 | 19 | 29

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | A. Coenzyme Q10 2400 mg/Day With Vitamin E 1200 IU/Day | B. Coenzyme Q10 1200 mg/Day With Vitamin E 1200 IU/Day | C. Placebo With Vitamin E 1200 IU/Day | Total
Number analyzed (Participants) | 196 | 201 | 203 | 600
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 113 | 113 | 133 | 359
  >=65 years | 83 | 88 | 70 | 241
Age Continuous [Mean (Standard Deviation); unit: years] | 62.8 (9.66) | 63.3 (9.83) | 61.3 (10.5) | 62.5 (10.03)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 68 | 62 | 73 | 203
  Male | 128 | 139 | 130 | 397
Region of Enrollment [Number; unit: participants]
  United States | 165 | 171 | 174 | 510
  Canada | 31 | 30 | 29 | 90

OUTCOME MEASURES:

1. Primary Outcome: Change in Unified Parkinson's Disease Rating Scale (UPDRS) (Total Score (Sum of Parts I, II and III Ranges From 0 to 176))
Description: Outcome is defined as change in total Unified Parkinson's Disease Rating Scale (UPDRS) between the baseline visit and month 16 or the time of sufficient disability to require dopaminergic therapy or study closure, whichever occurs first. The UPDRS score has three components, each consisting of questions answered on a 0-4 point scale. Part I assesses mentation, behavior and mood; Part II assesses activities of daily living in the week prior to the designated visit; and Part III assesses motor abilities at the time of the visit. A total of 31 items are included in Parts I, II and III. Each item will receive a score ranging from 0 to 4 where 0 represents the absence of impairment and 4 represents the highest degree of impairment. Total score ranges from 0-176.
Time Frame: Baseline to 16 months or the time of sufficient disability to require dopaminergic therapy or study closure, whichever occurs first
Population: Eligible research participants were assigned by randomization to one of three treatment groups: CoQ10 2400 mg/day, CoQ10 1200 mg/day or matching placebo. All participants also received 1200 IU of vitamin E daily.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | A. Coenzyme Q10 2400 mg/Day With Vitamin E 1200 IU/Day | B. Coenzyme Q10 1200 mg/Day With Vitamin E 1200 IU/Day | C. Placebo With Vitamin E 1200 IU/Day
Number analyzed (Participants) | 196 | 201 | 203
units on a scale | 8.01 (.63) | 7.50 (.62) | 6.92 (.63)
Statistical Analysis 1: Comparison: B. Coenzyme Q10 1200 mg/Day With Vitamin E 1200 IU/Day vs C. Placebo With Vitamin E 1200 IU/Day; ANCOVA is used with the change in total UPDRS of Coenzyme Q10 1200 mg/day arm compared to placebo group; Test type: Superiority or Other; p > 0.025, ANCOVA — The primary analysis compares each active treatment arm to the placebo arm. P-values for efficacy outcomes will be 2-sided, with a Bonferroni-adjusted significance level of .025 used to preserve the overall alpha level for the 2 comparisons at .05; Mean Difference (Net) = .59, 97.5% CI 2-sided [-1.33 to 2.51], Standard Error of Mean 0.85
Statistical Analysis 2: Comparison: A. Coenzyme Q10 2400 mg/Day With Vitamin E 1200 IU/Day vs C. Placebo With Vitamin E 1200 IU/Day; ANCOVA is used with the change in total UPDRS of Coenzyme Q10 2400 mg/day arm compared to placebo group; Test type: Superiority or Other; p > 0.025, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Net) = 1.09, 95% CI 2-sided [-0.85 to 3.03], Standard Error of Mean 0.86

2. Secondary Outcome: Change in Modified Schwab & England Independence Scale From Baseline to 16 Months
Description: This scale measures activities of daily living. This is an investigator and subject assessment of the subject's level of independence at all scheduled visits. The subject is scored on a percentage scale reflective of his/her ability to perform acts of daily living in relation to pre-Parkinson disease ability. Scores range in increments of 10%: 100% for normal (subject is completely independent; essentially normal) to 0% (vegetative functions such as swallowing, bladder and bowel functions are not functioning; bedridden).
Time Frame: as for outcome 1
Population: All participants were used in primary and secondary outcome analyses.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | A. Coenzyme Q10 2400 mg/Day With Vitamin E 1200 IU/Day | B. Coenzyme Q10 1200 mg/Day With Vitamin E 1200 IU/Day | C. Placebo With Vitamin E 1200 IU/Day
Number analyzed (Participants) | 196 | 201 | 203
units on a scale | -4.94 (.62) | -4.29 (.62) | -4.07 (.62)
Statistical Analysis 1: Comparison: B. Coenzyme Q10 1200 mg/Day With Vitamin E 1200 IU/Day vs C. Placebo With Vitamin E 1200 IU/Day; Change from Baseline Visit to 16-month visit on Modified Schwab & England will be analyzed using ANCOVA in the same way as for the primary outcome variable; Test type: Superiority or Other; p = 0.7943, ANCOVA — The primary analysis compares each active treatment arm to the placebo arm. P-Values for efficacy outcomes are 2-sided, with a Bonferroni-adjusted significance level of .025 used to preserve the overall alpha level for the 2 comparisons at .05; COCF is used for missing data and those lost to follow up. Outliers and non-compliant patients are assessed with scatter and residual plots and ITT; Mean Difference (Net) = -0.22, 97.5% CI 2-sided [-2.12 to 1.68], Standard Error of Mean 0.84
Statistical Analysis 2: Comparison: A. Coenzyme Q10 2400 mg/Day With Vitamin E 1200 IU/Day vs C. Placebo With Vitamin E 1200 IU/Day; Change from Baseline Visit to 16-month on Modified Schwab & England will be analyzed using ANCOVA in the same way as for the primary outcome variable; Test type: Superiority or Other; p = 0.306, ANCOVA — [p-value comment as in outcome 2, analysis 1]; [statistical method as in outcome 2, analysis 1]; Mean Difference (Net) = -0.87, 95% CI [-2.79 to 1.04], Standard Error of Mean 0.85

3. Secondary Outcome: Change in Modified Rankin Scale From Baseline to 16 Months
Description: The Modified Rankin Scale is a global functional health index with a strong accent on physical disability. Subjects are scored on a scale of 0 (no symptoms at all) to 5 (severe disability: bedridden incontinent, and requiring constant nursing care and attention.
Time Frame: as for outcome 1
Population: All participants were used in primary and secondary outcome analyses.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | A. Coenzyme Q10 2400 mg/Day With Vitamin E 1200 IU/Day | B. Coenzyme Q10 1200 mg/Day With Vitamin E 1200 IU/Day | C. Placebo With Vitamin E 1200 IU/Day
Number analyzed (Participants) | 196 | 201 | 203
units on a scale | .38 (.05) | .31 (.05) | .40 (.05)
Statistical Analysis 1: Comparison: B. Coenzyme Q10 1200 mg/Day With Vitamin E 1200 IU/Day vs C. Placebo With Vitamin E 1200 IU/Day; Change from Baseline Visit to 16-month visit on Modified Rankin Scale will be analyzed using ANCOVA in the same way as for the primary outcome variable; Test type: Superiority or Other; p < 0.1615, ANCOVA — [p-value comment as in outcome 2, analysis 1]; [statistical method as in outcome 2, analysis 1]; Mean Difference (Net) = -0.09, 97.5% CI 2-sided [-0.25 to 0.06], Standard Error of Mean 0.06
Statistical Analysis 2: Comparison: A. Coenzyme Q10 2400 mg/Day With Vitamin E 1200 IU/Day vs C. Placebo With Vitamin E 1200 IU/Day; Change from Baseline Visit to 16-month visit on Modified Rankin will be analyzed using ANCOVA in the same way as for the primary outcome variable; Test type: Superiority or Other; p = 0.7627, ANCOVA — [p-value comment as in outcome 2, analysis 1]; COCF is used for missing data and those lost to follow up. Outliers and non-compliant patients are assessed with scatter and residual plats and ITT; Mean Difference (Net) = -0.02, 95% CI 2-sided [-0.17 to 0.13], Standard Error of Mean 0.07

4. Secondary Outcome: Change in PD Quality of Life Scale From Baseline to 16 Months
Description: The subject will complete a questionnaire that will evaluate how Parkinson disease has affected their health and overall quality of life at each visit. The total quality of life scale measures a total of 33 aspects of quality of life. Each aspect is rated on scale of 0 (best outcome) to 4 (worst outcome). Total score range is 0-132. A higher score or increased score compared to a previous visit indicates a lowered quality of life.
Time Frame: as for outcome 1
Population: All participants were used in primary and secondary outcome analyses.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | A. Coenzyme Q10 2400 mg/Day With Vitamin E 1200 IU/Day | B. Coenzyme Q10 1200 mg/Day With Vitamin E 1200 IU/Day | C. Placebo With Vitamin E 1200 IU/Day
Number analyzed (Participants) | 196 | 201 | 203
units on a scale | 5.06 (.89) | 6.12 (.87) | 5.57 (.89)
Statistical Analysis 1: Comparison: B. Coenzyme Q10 1200 mg/Day With Vitamin E 1200 IU/Day vs C. Placebo With Vitamin E 1200 IU/Day; Change from Baseline Visit to 16-month visit on PD Quality of Life Scale will be analyzed using ANCOVA in the same way as for the primary outcome variable; Test type: Superiority or Other; p = 0.6383, ANCOVA — [p-value comment as in outcome 2, analysis 1]; [statistical method as in outcome 2, analysis 1]; Mean Difference (Net) = 0.6383, 97.5% CI 2-sided [-2.10 to 3.21], Standard Error of Mean 1.18
Statistical Analysis 2: Comparison: A. Coenzyme Q10 2400 mg/Day With Vitamin E 1200 IU/Day vs C. Placebo With Vitamin E 1200 IU/Day; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.667, ANCOVA — [p-value comment as in outcome 2, analysis 1]; [statistical method as in outcome 2, analysis 1]; Mean Difference (Net) = -0.51, 95% CI 2-sided [-3.20 to 2.17], Standard Error of Mean 1.19

5. Secondary Outcome: Change in Symbol Digit Modalities Test From Baseline to 16 Months
Description: The Symbol Digit Modalities Test screens cognitive impairment by using a simple substitution tasks that individuals with normal functioning can easily perform. The test score range is from 0(worst outcome) to 110 (best outcome).
Time Frame: as for outcome 1
Population: All participants were used in primary and secondary outcome analyses.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | A. Coenzyme Q10 2400 mg/Day With Vitamin E 1200 IU/Day | B. Coenzyme Q10 1200 mg/Day With Vitamin E 1200 IU/Day | C. Placebo With Vitamin E 1200 IU/Day
Number analyzed (Participants) | 196 | 201 | 203
units on a scale | -3.36 (1.40) | -0.49 (1.39) | -3.02 (1.48)
Statistical Analysis 1: Comparison: B. Coenzyme Q10 1200 mg/Day With Vitamin E 1200 IU/Day vs C. Placebo With Vitamin E 1200 IU/Day; Change from Baseline Visit to 16-month visit on Symbol Digit Modalities Test will be analyzed using ANCOVA in the same way as for the primary outcome variable; Test type: Superiority or Other; p = 0.671, ANCOVA — [p-value comment as in outcome 2, analysis 1]; [statistical method as in outcome 2, analysis 1]; Mean Difference (Net) = 0.49, 97.5% CI 2-sided [-2.09 to 3.06], Standard Error of Mean 1.14
Statistical Analysis 2: Comparison: A. Coenzyme Q10 2400 mg/Day With Vitamin E 1200 IU/Day vs C. Placebo With Vitamin E 1200 IU/Day; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; p = 0.671, ANCOVA — [p-value comment as in outcome 2, analysis 1]; [statistical method as in outcome 2, analysis 1]; Mean Difference (Net) = -0.74, 95% CI 2-sided [-3.34 to 1.87], Standard Error of Mean 1.16

6. Secondary Outcome: Change in Hoehn & Yahr Score From Baseline to 16 Months
Description: The Modified Hoehn and Yahr Scale is an 8-level Parkinson disease staging instrument. The investigator will assess disease stage at each level. The disease stages range from the best outcome of 0 (no signs of disease) to the worst outcome of 5 (wheelchair bound or bedridden unless aided).
Time Frame: as for outcome 1
Population: All participants were used in primary and secondary outcome analyses.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | A. Coenzyme Q10 2400 mg/Day With Vitamin E 1200 IU/Day | B. Coenzyme Q10 1200 mg/Day With Vitamin E 1200 IU/Day | C. Placebo With Vitamin E 1200 IU/Day
Number analyzed (Participants) | 196 | 201 | 203
units on a scale | .21 (0.03) | .20 (0.03) | .16 (0.03)
Statistical Analysis 1: Comparison: B. Coenzyme Q10 1200 mg/Day With Vitamin E 1200 IU/Day vs C. Placebo With Vitamin E 1200 IU/Day; Change from Baseline Visit to 16-month visit on Hoehn & Yahr Score will be analyzed using ANCOVA in the same way as for the primary outcome variable; Test type: Superiority or Other; p = 0.3445, ANCOVA — [p-value comment as in outcome 2, analysis 1]; [statistical method as in outcome 2, analysis 1]; Mean Difference (Net) = 0.04, 97.5% CI 2-sided [-0.04 to 0.13], Standard Error of Mean 0.04
Statistical Analysis 2: Comparison: A. Coenzyme Q10 2400 mg/Day With Vitamin E 1200 IU/Day vs C. Placebo With Vitamin E 1200 IU/Day; Change from Baseline visit to 16-month visit on Hoehn & Yahr will be analyzed using ANCOVA in the same way as for the primary outcome variable; Test type: Superiority or Other; p = .239, ANCOVA — The primary analysis compares each active treatment arm to the placebo arm. P-Values for efficacy outcomes are 2-sided. with a Bonferroni-adjustd significance level of .025 used to preserve the overall alpha level for the 2 comparisons at .05; COCF is used for missing data and those lost to follow up. Outliers and non-compliant patients are assess with scatter and residual plots and ITT; Mean Difference (Net) = 0.04, 95% CI [-0.04 to 0.14], Standard Error of Mean 0.05

7. Secondary Outcome: CoQ10 Levels in Plasma
Description: Based on samples analyzed to date
Time Frame: Baseline, 1, 8 and 16 months or the time of sufficient disability to require dopaminergic therapy or study closure, whichever occurs first
Population: All participants have been included and data is based on samples analyzed to date.
Measure: Mean (Standard Deviation); unit: ug/ml
Arm/Group | A. Coenzyme Q10 2400 mg/Day With Vitamin E 1200 IU/Day | B. Coenzyme Q10 1200 mg/Day With Vitamin E 1200 IU/Day | C. Placebo With Vitamin E 1200 IU/Day
Number analyzed (Participants) | 196 | 201 | 203
ug/ml
  1 month visit | 3.55 (1.83) | 2.57 (1.29) | .75 (.36)
  8 month visit | 3.32 (1.93) | 2.67 (1.33) | 1.07 (.83)
  16 month visit | 2.88 (2.02) | 2.17 (1.18) | .63 (.27)
Statistical Analysis 1: Comparison: A. Coenzyme Q10 2400 mg/Day With Vitamin E 1200 IU/Day vs B. Coenzyme Q10 1200 mg/Day With Vitamin E 1200 IU/Day vs C. Placebo With Vitamin E 1200 IU/Day; The analysis will be using the actual change of plasma levels of CoQ10(from final visit to baseline) as predictors of UPDRS worsening. Correlation of UPDRS worsening with plasma levels of CoQ10 will be calculated for all treatment groups; Test type: Superiority or Other; p = 0.0577, ANOVA; The ANOVA is using UPDRS worsening as outcome, Change of CoQ10 level as predictor, adjusting for site and baseline UPDRS score; Slope = 0.536, 95% CI 2-sided [-0.018 to 1.091], Standard Error of Mean 0.282
Statistical Analysis 2: Comparison: A. Coenzyme Q10 2400 mg/Day With Vitamin E 1200 IU/Day; The analysis will be using the actual change of plasma levels of CoQ10(from final to baseline) as predictors of UPDRS worsening. Correlation of UPDRS worsening with plasma levels of CoQ10 will be calculated for the treatment group of Coenzyme Q10 2400 mg/day; Test type: Superiority or Other; p = 0.5889, ANOVA; [statistical method as in outcome 7, analysis 1]; Slope = 0.245, 95% CI 2-sided [-0.647 to 1.136], Standard Error of Mean 0.451
Statistical Analysis 3: Comparison: B. Coenzyme Q10 1200 mg/Day With Vitamin E 1200 IU/Day; The analysis will be using the actual change of plasma levels of CoQ10(from final to baseline) as predictors of UPDRS worsening. Correlation of UPDRS worsening with plasma levels of CoQ10 will be calculated for the treatment group of Coenzyme Q10 1200 mg/day; Test type: Superiority or Other; p = 0.3006, ANOVA; [statistical method as in outcome 7, analysis 1]; Slope = 0.631, 95% CI 2-sided [-0.569 to 1.831], Standard Error of Mean 0.608
Statistical Analysis 4: Comparison: C. Placebo With Vitamin E 1200 IU/Day; The analysis will be using the actual change of plasma levels of CoQ10(from final to baseline) as predictors of UPDRS worsening. Correlation of UPDRS worsening with plasma levels of CoQ10 will be calculated for the placebo group; Test type: Superiority or Other; p = 0.096, ANOVA; [statistical method as in outcome 7, analysis 1]; Slope = 2.126, 95% CI 2-sided [-0.382 to 4.633], Standard Error of Mean 1.269

8. Secondary Outcome: Adverse Experiences: Back Pain
Description: Number of participants with back pain
Time Frame: Over 16 months (Screening, Baseline, 1, 4, 8, 12 and 16 month visits)
Population: All participants were used in primary and secondary outcome analysis.
Measure: Number; unit: participants
Arm/Group | A. Coenzyme Q10 2400 mg/Day With Vitamin E 1200 IU/Day | B. Coenzyme Q10 1200 mg/Day With Vitamin E 1200 IU/Day | C. Placebo With Vitamin E 1200 IU/Day
Number analyzed (Participants) | 196 | 201 | 203
participants | 9 | 13 | 9
Statistical Analysis 1: Comparison: A. Coenzyme Q10 2400 mg/Day With Vitamin E 1200 IU/Day vs B. Coenzyme Q10 1200 mg/Day With Vitamin E 1200 IU/Day vs C. Placebo With Vitamin E 1200 IU/Day; All adverse experiences were tabulated by treatment group, severity and perceived relationship to study medication. Fisher's exact test was used to compare active treatment arms to the placebo arm with regard to the proportion of subjects experiencing a particular adverse experience; Test type: Superiority or Other; p < 0.05, Fisher Exact; Odds Ratio (OR) = 1.26, 95% CI 2-sided [0.57 to 2.80], Standard Error of Mean 0.0199 — Odds ratio >1 indicates a higher frequency in active treatment group

9. Secondary Outcome: Adverse Experiences: Constipation
Description: Number of participants with constipation
Time Frame: Over 16 months (Screening, Baseline, 1, 4, 8, 12 and 16 month visits)
Population: All participants were used in primary and secondary outcome analysis.
Measure: Number; unit: participants
Arm/Group | A. Coenzyme Q10 2400 mg/Day With Vitamin E 1200 IU/Day | B. Coenzyme Q10 1200 mg/Day With Vitamin E 1200 IU/Day | C. Placebo With Vitamin E 1200 IU/Day
Number analyzed (Participants) | 196 | 201 | 203
participants | 7 | 13 | 7
Statistical Analysis 1: Comparison: A. Coenzyme Q10 2400 mg/Day With Vitamin E 1200 IU/Day vs B. Coenzyme Q10 1200 mg/Day With Vitamin E 1200 IU/Day vs C. Placebo With Vitamin E 1200 IU/Day; All adverse experiences were tabulated by treatment group, severity and perceived relationship to study medication. Fisher's exact test was used to compare active treatment arms to the placebo arm with regard to the proportion of subject experiencing a particular adverse experience; Test type: Superiority or Other; p < 0.05, Fisher Exact; Odds Ratio (OR) = 1.49, 95% CI 2-sided [0.62 to 3.57], Standard Error of Mean 0.0198 — Odds ratio >1 indicates a higher frequency in active treatment group

10. Secondary Outcome: Adverse Experiences: Insomnia
Description: Number of participants with insomnia
Time Frame: Over 16 months (Screening, Baseline, 1, 4, 8, 12 and 16 month visits)
Population: All participants were used in primary and secondary outcome analysis.
Measure: Number; unit: participants
Arm/Group | A. Coenzyme Q10 2400 mg/Day With Vitamin E 1200 IU/Day | B. Coenzyme Q10 1200 mg/Day With Vitamin E 1200 IU/Day | C. Placebo With Vitamin E 1200 IU/Day
Number analyzed (Participants) | 196 | 201 | 203
participants | 6 | 13 | 6
Statistical Analysis 1: Comparison: A. Coenzyme Q10 2400 mg/Day With Vitamin E 1200 IU/Day vs B. Coenzyme Q10 1200 mg/Day With Vitamin E 1200 IU/Day vs C. Placebo With Vitamin E 1200 IU/Day; [analysis description as in outcome 8, analysis 1]; Test type: Superiority or Other; p < 0.05, Fisher Exact; Odds Ratio (OR) = 1.65, 95% CI 2-sided [0.65 to 4.20], Standard Error of Mean 0.0198 — Odds ratio >1 indicates a higher frequency in active treatment group

11. Secondary Outcome: Adverse Experiences: Anxiety
Description: Number of participants with anxiety
Time Frame: Over 16 months (Screening, Baseline, 1, 4, 8, 12 and 16 month visits)
Population: All participants were used in primary and secondary outcome analysis.
Measure: Number; unit: participants
Arm/Group | A. Coenzyme Q10 2400 mg/Day With Vitamin E 1200 IU/Day | B. Coenzyme Q10 1200 mg/Day With Vitamin E 1200 IU/Day | C. Placebo With Vitamin E 1200 IU/Day
Number analyzed (Participants) | 196 | 201 | 203
participants | 12 | 13 | 14
Statistical Analysis 1: Comparison: A. Coenzyme Q10 2400 mg/Day With Vitamin E 1200 IU/Day vs B. Coenzyme Q10 1200 mg/Day With Vitamin E 1200 IU/Day vs C. Placebo With Vitamin E 1200 IU/Day; [analysis description as in outcome 8, analysis 1]; Test type: Superiority or Other; p < 0.05, ANCOVA; Odds Ratio (OR) = 0.91, 95% CI 2-sided [0.46 to 1.79], Standard Error of Mean 0.0200 — Odds ratio >1 indicates a higher frequency in active treatment group

12. Secondary Outcome: Adverse Experiences: Tremor
Description: Number of participants with tremor
Time Frame: Over 16 months (Screening, Baseline, 1, 4, 8, 12 and 16 month visits)
Population: All participants were used in primary and secondary outcome analysis.
Measure: Number; unit: participants
Arm/Group | A. Coenzyme Q10 2400 mg/Day With Vitamin E 1200 IU/Day | B. Coenzyme Q10 1200 mg/Day With Vitamin E 1200 IU/Day | C. Placebo With Vitamin E 1200 IU/Day
Number analyzed (Participants) | 196 | 201 | 203
participants | 10 | 13 | 8
Statistical Analysis 1: Comparison: A. Coenzyme Q10 2400 mg/Day With Vitamin E 1200 IU/Day vs B. Coenzyme Q10 1200 mg/Day With Vitamin E 1200 IU/Day vs C. Placebo With Vitamin E 1200 IU/Day; [analysis description as in outcome 8, analysis 1]; Test type: Superiority or Other; p < 0.05, Fisher Exact; Odds Ratio (OR) = 1.50, 95% CI 2-sided [0.66 to 3.41], Standard Error of Mean 0.0199 — Odds ratio >1 indicates a higher frequency in active treatment group

13. Secondary Outcome: Adverse Experiences: Nasopharyngitis
Description: Number of participants with nasopharyngitis
Time Frame: Over 16 months (Screening, Baseline, 1, 4, 8, 12 and 16 month visits)
Population: All participants were used in primary and secondary outcome analysis.
Measure: Number; unit: participants
Arm/Group | A. Coenzyme Q10 2400 mg/Day With Vitamin E 1200 IU/Day | B. Coenzyme Q10 1200 mg/Day With Vitamin E 1200 IU/Day | C. Placebo With Vitamin E 1200 IU/Day
Number analyzed (Participants) | 196 | 201 | 203
participants | 7 | 9 | 3
Statistical Analysis 1: Comparison: A. Coenzyme Q10 2400 mg/Day With Vitamin E 1200 IU/Day vs B. Coenzyme Q10 1200 mg/Day With Vitamin E 1200 IU/Day vs C. Placebo With Vitamin E 1200 IU/Day; [analysis description as in outcome 8, analysis 1]; Test type: Superiority or Other; p < 0.05, Fisher Exact; Odds Ratio (OR) = 2.80, 95% CI 2-sided [0.81 to 9.72], Standard Error of Mean 0.0197 — Odds ratio >1 indicates a higher frequency in active treatment group

14. Secondary Outcome: Adverse Experiences: Diarrhoea
Description: Number of participants with diarrhoea
Time Frame: Over 16 months (Screening, Baseline, 1, 4, 8, 12 and 16 month visits)
Population: All participants were used in primary and secondary outcome analysis.
Measure: Number; unit: participants
Arm/Group | A. Coenzyme Q10 2400 mg/Day With Vitamin E 1200 IU/Day | B. Coenzyme Q10 1200 mg/Day With Vitamin E 1200 IU/Day | C. Placebo With Vitamin E 1200 IU/Day
Number analyzed (Participants) | 196 | 201 | 203
participants | 6 | 9 | 11
Statistical Analysis 1: Comparison: A. Coenzyme Q10 2400 mg/Day With Vitamin E 1200 IU/Day vs B. Coenzyme Q10 1200 mg/Day With Vitamin E 1200 IU/Day vs C. Placebo With Vitamin E 1200 IU/Day; [analysis description as in outcome 8, analysis 1]; Test type: Superiority or Other; p < 0.05, Fisher Exact; Odds Ratio (OR) = 0.69, 95% CI 2-sided [0.31 to 1.52], Standard Error of Mean 0.0197 — Odds ratio >1 indicates a higher frequency in active treatment group

15. Secondary Outcome: Adverse Experiences: Headache
Description: Number of participants with headache
Time Frame: Over 16 months (Screening, Baseline, 1, 4, 8, 12 and 16 month visits)
Population: All participants were used in primary and secondary outcome analysis.
Measure: Number; unit: participants
Arm/Group | A. Coenzyme Q10 2400 mg/Day With Vitamin E 1200 IU/Day | B. Coenzyme Q10 1200 mg/Day With Vitamin E 1200 IU/Day | C. Placebo With Vitamin E 1200 IU/Day
Number analyzed (Participants) | 196 | 201 | 203
participants | 9 | 8 | 11
Statistical Analysis 1: Comparison: A. Coenzyme Q10 2400 mg/Day With Vitamin E 1200 IU/Day vs B. Coenzyme Q10 1200 mg/Day With Vitamin E 1200 IU/Day vs C. Placebo With Vitamin E 1200 IU/Day; [analysis description as in outcome 8, analysis 1]; Test type: Superiority or Other; p < 0.05, Fisher Exact; Odds Ratio (OR) = 0.78, 95% CI 2-sided [0.36 to 1.70], Standard Error of Mean 0.0197 — Odds ratio >1 indicates a higher frequency in active treatment group

16. Secondary Outcome: Adverse Experiences: Urinary Tract Infection
Description: Number of patients with urinary tract infections
Time Frame: Over 16 months (Screening, Baseline, 1, 4, 8, 12 and 16 month visits)
Population: All participants were used in primary and secondary outcome analysis.
Measure: Number; unit: participants
Arm/Group | A. Coenzyme Q10 2400 mg/Day With Vitamin E 1200 IU/Day | B. Coenzyme Q10 1200 mg/Day With Vitamin E 1200 IU/Day | C. Placebo With Vitamin E 1200 IU/Day
Number analyzed (Participants) | 196 | 201 | 203
participants | 6 | 8 | 3
Statistical Analysis 1: Comparison: A. Coenzyme Q10 2400 mg/Day With Vitamin E 1200 IU/Day vs B. Coenzyme Q10 1200 mg/Day With Vitamin E 1200 IU/Day vs C. Placebo With Vitamin E 1200 IU/Day; [analysis description as in outcome 8, analysis 1]; Test type: Superiority or Other; p < 0.05, Fisher Exact; Odds Ratio (OR) = 2.44, 95% CI 2-sided [0.69 to 8.58], Standard Error of Mean 0.0197 — Odds ratio >1 indicates a higher frequency in active treatment group

17. Secondary Outcome: Adverse Experiences: Nausea
Description: Number of participants with nausea
Time Frame: Over 16 months (Screening, Baseline, 1, 4, 8, 12 and 16 month visits)
Population: All participants were used in primary and secondary outcome analysis.
Measure: Number; unit: participants
Arm/Group | A. Coenzyme Q10 2400 mg/Day With Vitamin E 1200 IU/Day | B. Coenzyme Q10 1200 mg/Day With Vitamin E 1200 IU/Day | C. Placebo With Vitamin E 1200 IU/Day
Number analyzed (Participants) | 196 | 201 | 203
participants | 7 | 7 | 10
Statistical Analysis 1: Comparison: A. Coenzyme Q10 2400 mg/Day With Vitamin E 1200 IU/Day vs B. Coenzyme Q10 1200 mg/Day With Vitamin E 1200 IU/Day vs C. Placebo With Vitamin E 1200 IU/Day; [analysis description as in outcome 8, analysis 1]; Test type: Superiority or Other; p < 0.05, Fisher Exact; Odds Ratio (OR) = 0.71, 95% CI 2-sided [0.31 to 1.62], Standard Error of Mean 0.0197 — Odds ratio >1 indicates a higher frequency in active treatment group

18. Secondary Outcome: Adverse Experiences: Hypertension
Description: Number of participants with hypertension
Time Frame: Over 16 months (Screening, Baseline, 1, 4, 8, 12 and 16 month visits)
Population: All participants were used in primary and secondary outcome analysis.
Measure: Number; unit: participants
Arm/Group | A. Coenzyme Q10 2400 mg/Day With Vitamin E 1200 IU/Day | B. Coenzyme Q10 1200 mg/Day With Vitamin E 1200 IU/Day | C. Placebo With Vitamin E 1200 IU/Day
Number analyzed (Participants) | 196 | 201 | 203
participants | 5 | 7 | 0
Statistical Analysis 1: Comparison: A. Coenzyme Q10 2400 mg/Day With Vitamin E 1200 IU/Day vs B. Coenzyme Q10 1200 mg/Day With Vitamin E 1200 IU/Day vs C. Placebo With Vitamin E 1200 IU/Day; [analysis description as in outcome 8, analysis 1]; Test type: Superiority or Other; p < 0.05, Fisher Exact; Odds Ratio (OR) = 9999.98, 95% CI 2-sided [2.77 to 9999.99], Standard Error of Mean 0.0196 — Odds ratio >1 indicates a higher frequency in active treatment group

19. Secondary Outcome: Adverse Experiences: Depression
Description: Number of participants with depression
Time Frame: Over 16 months (Screening, Baseline, 1, 4, 8, 12 and 16 month visits)
Population: All participants were used in primary and secondary outcome analysis.
Measure: Number; unit: participants
Arm/Group | A. Coenzyme Q10 2400 mg/Day With Vitamin E 1200 IU/Day | B. Coenzyme Q10 1200 mg/Day With Vitamin E 1200 IU/Day | C. Placebo With Vitamin E 1200 IU/Day
Number analyzed (Participants) | 196 | 201 | 203
participants | 9 | 6 | 14
Statistical Analysis 1: Comparison: A. Coenzyme Q10 2400 mg/Day With Vitamin E 1200 IU/Day vs B. Coenzyme Q10 1200 mg/Day With Vitamin E 1200 IU/Day vs C. Placebo With Vitamin E 1200 IU/Day; [analysis description as in outcome 8, analysis 1]; Test type: Superiority or Other; p < 0.05, Fisher Exact; Odds Ratio (OR) = 0.53, 95% CI 2-sided [0.25 to 1.12], Standard Error of Mean 0.0197 — Odds ration >1 indicates a higher frequency in active treatment group

20. Secondary Outcome: Adverse Experiences: Constipation: Moderate/Severe
Description: Number of participants with moderate/severe constipation
Time Frame: Over 16 months (Screening, Baseline, 1, 4, 8, 12 and 16 month visits)
Population: All participants were used in primary and secondary outcome analysis.
Measure: Number; unit: participants
Arm/Group | A. Coenzyme Q10 2400 mg/Day With Vitamin E 1200 IU/Day | B. Coenzyme Q10 1200 mg/Day With Vitamin E 1200 IU/Day | C. Placebo With Vitamin E 1200 IU/Day
Number analyzed (Participants) | 196 | 201 | 203
participants | 3 | 10 | 3
Statistical Analysis 1: Comparison: A. Coenzyme Q10 2400 mg/Day With Vitamin E 1200 IU/Day vs B. Coenzyme Q10 1200 mg/Day With Vitamin E 1200 IU/Day vs C. Placebo With Vitamin E 1200 IU/Day; [analysis description as in outcome 8, analysis 1]; Test type: Superiority or Other; p < 0.05, Fisher Exact; Odds Ratio (OR) = 2.26, 95% CI 2-sided [0.64 to 8.01], Standard Error of Mean 0.0196 — Odds ratio >1 indicates a higher frequency in active treatment group

21. Secondary Outcome: Adverse Experiences: Anxiety: Moderate/Severe
Description: Number of participants with moderate/severe anxiety
Time Frame: Over 16 months (Screening, Baseline, 1, 4, 8, 12 and 16 month visits)
Population: All participants were used in primary and secondary outcome analysis.
Measure: Number; unit: participants
Arm/Group | A. Coenzyme Q10 2400 mg/Day With Vitamin E 1200 IU/Day | B. Coenzyme Q10 1200 mg/Day With Vitamin E 1200 IU/Day | C. Placebo With Vitamin E 1200 IU/Day
Number analyzed (Participants) | 196 | 201 | 203
participants | 9 | 9 | 7
Statistical Analysis 1: Comparison: A. Coenzyme Q10 2400 mg/Day With Vitamin E 1200 IU/Day vs B. Coenzyme Q10 1200 mg/Day With Vitamin E 1200 IU/Day vs C. Placebo With Vitamin E 1200 IU/Day; [analysis description as in outcome 8, analysis 1]; Test type: Superiority or Other; p < 0.05, Fisher Exact; Odds Ratio (OR) = 1.33, 95% CI 2-sided [0.55 to 3.24], Standard Error of Mean 0.0198 — Odds ratio of >1 indicates a higher frequency in active treatment group

22. Secondary Outcome: Adverse Experiences: Back Pain: Moderate/Severe
Description: Number of participants with moderate/severe back pain
Time Frame: Over 16 months (Screening, Baseline, 1, 4, 8, 12 and 16 month visits)
Population: All participants were used in primary and secondary outcome analysis.
Measure: Number; unit: participants
Arm/Group | A. Coenzyme Q10 2400 mg/Day With Vitamin E 1200 IU/Day | B. Coenzyme Q10 1200 mg/Day With Vitamin E 1200 IU/Day | C. Placebo With Vitamin E 1200 IU/Day
Number analyzed (Participants) | 196 | 201 | 203
participants | 7 | 9 | 7
Statistical Analysis 1: Comparison: A. Coenzyme Q10 2400 mg/Day With Vitamin E 1200 IU/Day vs B. Coenzyme Q10 1200 mg/Day With Vitamin E 1200 IU/Day vs C. Placebo With Vitamin E 1200 IU/Day; [analysis description as in outcome 8, analysis 1]; Test type: Superiority or Other; p < 0.05, Fisher Exact; Odds Ratio (OR) = 9999.98, 95% CI 2-sided [0.48 to 9999.99], Standard Error of Mean 0.0197 — Odds ratio >1 indicates a higher frequency in active treatment group

23. Secondary Outcome: Adverse Experiences: Insomnia: Moderate/Severe
Description: Number of participants with moderate/severe insomnia
Time Frame: Over 16 months (Screening, Baseline, 1, 4, 8, 12 and 16 month visits)
Population: All participants were used in primary and secondary outcome analysis.
Measure: Number; unit: participants
Arm/Group | A. Coenzyme Q10 2400 mg/Day With Vitamin E 1200 IU/Day | B. Coenzyme Q10 1200 mg/Day With Vitamin E 1200 IU/Day | C. Placebo With Vitamin E 1200 IU/Day
Number analyzed (Participants) | 196 | 201 | 203
participants | 2 | 9 | 0
Statistical Analysis 1: Comparison: A. Coenzyme Q10 2400 mg/Day With Vitamin E 1200 IU/Day vs B. Coenzyme Q10 1200 mg/Day With Vitamin E 1200 IU/Day vs C. Placebo With Vitamin E 1200 IU/Day; [analysis description as in outcome 8, analysis 1]; Test type: Superiority or Other; p < 0.05, Fisher Exact; Odds Ratio (OR) = 9999.98, 95% CI 2-sided [2.51 to 9999.99], Standard Error of Mean 0.0196 — Odds ratio >1 indicates a higher frequency in active treatment group

ADVERSE EVENTS:
Time Frame: Adverse events data were collected for a period of 2 years and 7 months.
Arm/Group | A. Coenzyme Q10 2400 mg/Day With Vitamin E 1200 IU/Day | B. Coenzyme Q10 1200 mg/Day With Vitamin E 1200 IU/Day | C. Placebo With Vitamin E 1200 IU/Day
Serious Adverse Events (participants affected / at risk) | 7/196 | 13/201 | 13/203
Other Adverse Events (participants affected / at risk) | 106/196 | 113/201 | 108/203
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | A. Coenzyme Q10 2400 mg/Day With Vitamin E 1200 IU/Day (N=196) | B. Coenzyme Q10 1200 mg/Day With Vitamin E 1200 IU/Day (N=201) | C. Placebo With Vitamin E 1200 IU/Day (N=203)
Cardiac catheterization (Surgical and medical procedures) | 1 (1) | 0/0 (0) | 1 (1)
Gastero-intestinal bleed (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Multiple myeloma (General disorders) | 1 (1) | 0 (0) | 0 (0)
Prostatitis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Pacemaker battery replacement (Surgical and medical procedures) | 2 (2) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Cervical radiculopathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Back pain (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Bowel obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Vertigo (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Accident with fractures (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1)
Total knee replacement (Surgical and medical procedures) | 0 (0) | 1 (2) | 1 (1)
Gastric banding (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Chest pain (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Pelvic floor dysfunction (Reproductive system and breast disorders) | 0/68 (0) | 1/62 (1) | 0/73 (0)
Spinal stenosis (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Prostate cancer progression (Renal and urinary disorders) | 1/128 (1) | 0/139 (0) | 0/130 (0)
Breast cancer (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Pulmonary embolism (General disorders) | 0 (0) | 1 (1) | 0 (0)
Benign prostatic hypertrophy (Renal and urinary disorders) | 0/128 (0) | 0/139 (0) | 1/130 (1)
Pneumonia (General disorders) | 0 (0) | 0 (0) | 2 (2)
Transurethral resection of the prostate (Surgical and medical procedures) | 0/128 (0) | 1/139 (1) | 0/130 (0)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Sudden death (General disorders) | 0 (0) | 1 (1) | 0 (0)
Dental infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Hypersensitivity pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) | 0 (0)
Colon cancer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Dehydration (General disorders) | 0 (0) | 0 (0) | 1 (2)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Subarachnoid hemorrhage (General disorders) | 0 (0) | 0 (0) | 0 (0)
Accident with fractures and head trauma (General disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | A. Coenzyme Q10 2400 mg/Day With Vitamin E 1200 IU/Day (N=196) | B. Coenzyme Q10 1200 mg/Day With Vitamin E 1200 IU/Day (N=201) | C. Placebo With Vitamin E 1200 IU/Day (N=203)
Back pain (Nervous system disorders) | 9 (9) | 13 (13) | 9 (9)
Constipation (Gastrointestinal disorders) | 7 (7) | 13 (13) | 7 (7)
Insomnia (General disorders) | 6 (6) | 13 (13) | 6 (6)
Anxiety (Psychiatric disorders) | 12 (12) | 13 (13) | 14 (14)
Tremor (Nervous system disorders) | 10 (10) | 13 (13) | 8 (8)
Nasopharyngitis (General disorders) | 7 (7) | 9 (9) | 3 (3)
Diarrhea (Gastrointestinal disorders) | 6 (6) | 9 (9) | 11 (11)
Headache (General disorders) | 9 (9) | 8 (8) | 11 (11)
Urinary tract infection (Renal and urinary disorders) | 6 (6) | 8 (8) | 3 (3)
Nausea (Gastrointestinal disorders) | 7 (7) | 7 (7) | 10 (10)
Hypertension (Vascular disorders) | 5 (5) | 7 (7) | 0 (0)
Depression (Psychiatric disorders) | 9 (9) | 6 (6) | 14 (14)
Dizziness (Nervous system disorders) | 7 (7) | 6 (6) | 5 (5)
Fall (Injury, poisoning and procedural complications) | 6 (6) | 6 (6) | 7 (7)

LIMITATIONS AND CAVEATS:
The planned interim analysis for futility based on the first 300 subjects has reached the pre-specified termination criterion.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No